CLINICAL TRIAL: NCT05947578
Title: A Phase 1, Open-Label, Prospective, Dose-finding Clinical Trial for Evaluation of Safety and Tolerability of Intramuscular Injections of CLZ-2002 for the Treatment of Subjects With Charcot-Marie-Tooth Type 1(CMT 1)
Brief Title: The Safety and Tolerability of CLZ-2002 in Patients With Charcot-Marie Tooth Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellatoz Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLZ-CMT-101
Record Dates: First submitted 2023-06-16; First posted 2023-07-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2023-06

CONDITIONS: Charcot Marie Tooth Disease, Type 1
Keywords: Charcot-Marie-Tooth Disease; CMT1; Cell therapy; Tonsillar mesenchymal stem cells (T-MSC); Neuronal Regeneration Promoting Cells; Schwann cell-like cells
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Intervention Model Description: Dose group A (Low dose) Dose group B (Mid dose) Dose group C (High dose)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLZ-2002 (Experimental): CLZ-2002 injection is intramuscular in lower limbs on Day 1.
  Interventions: Drug: CLZ-2002

INTERVENTIONS:
Drug: CLZ-2002 — Low dose group (6×10^6 cells), Mid dose group (12×10^6 cells), High dose group (24×10^6 cells)
  Other Names: Allogeneic tonsillar mesenchymal stem cell-derived schwann cell like cells

SUMMARY:
A Phase 1, Open-Label, Prospective, Dose-finding Clinical Trial for Evaluation of Safety and Tolerability of Intramuscular Injections of CLZ-2002 for the Treatment of Subjects with Charcot-Marie-Tooth type 1(CMT 1)

DETAILED DESCRIPTION:
This study is the First In Human (FIH) clinical trial for evaluating the safety and tolerability of IM injections of CLZ-2002 in patients with Charcot-Marie-Tooth disease (CMT) Type 1.

CLZ-2002 is the allogeneic mesenchymal stem cell-derived Neuronal Regeneration Promoting Cells. These cells are Schwann cell-like cells differentiated from tonsillar mesenchymal stem cells. CLZ-2002 helps the remyelination of the damaged peripheral nerves by restoring the myelin sheaths. It also induces the nerve regeneration and myelination pathways in the sciatic nerve and restores abnormal muscle tissues in Charcot-Marie-Tooth disease type 1 (CMT1).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older
* Subjects with a proven diagnosis of Charcot-Marie-Tooth disease type 1 at the time of screening visit
* Subjects who have muscle weakness in at least foot dorsiflexion (clinical assessment) at the time of screening visit
* Subjects with a CMT neuropathy score (CMTNS-v2) of 2 or more and 30 or fewer points at the time of screening visit
* Subjects who can understand and are willing to sign a written informed consent document are willing to comply with all study procedures and schedule visits.

Exclusion Criteria:

* Subjects who have any other neuromuscular diseases
* Subjects who have undergone upper and lower limb bone surgery within six months before screening visit
* Subjects who have concerns about muscle strength measurements due to the previous surgery
* Subjects who have severe active infection including severe/purulent cellulitis at the injection sites at screening visit
* Subjects who have a history of hospitalization due to hypersensitivity to antihistamines or allergy or hypersensitivity to certain substances such as food or drugs
* Subjects who have a history of unstable cardiovascular disease defined by the presence of myocardial infarction (STEMI or NSTEMI) within 6 months before the screening or the presence of unstable angina pectoris (in the case of increased frequency of symptoms, increased severity, or signs of prolonged symptoms at moderate activity or rest)
* Subjects who have a history of a transient ischemic attack (TIA) or stroke within 6 months before screening visit
* Subjects who have a positive HIV antibody test, hepatitis B antigen, or hepatitis C antibody test result
* Subjects who have a history of malignant tumors within 5 years before screening visit
* Subjects who have received systemic steroids (inhaled steroids are allowed), immunotherapy, or cytotoxic therapy within 14 days before screening, or who are expected to receive such treatment during the study period
* Subjects who have participated in other clinical trials within 30 days before screening visit
* Pregnant and lactating women or women of childbearing potential and men who plan a pregnancy or are unwilling to use adequate birth control methods& until 30 days after the end of drug administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of intramuscular (IM) injections of CLZ-2002 in Participants | Day 1 (visit 2) to Week 24 (visit 6)
  Frequency and percentage of treatment-emergent adverse events (TEAEs) and serious adverse events after injection through laboratory tests, physical examinations, vital signs, and electrocardiogram measurements conducted during the clinical trial.

SECONDARY OUTCOMES:
Changes from baseline in the disease severity of CMTNS-v2 score at Weeks 4, 12, and 24. | Weeks 4, 12 and 24
  The range of CMTNS-v2 (Charcot Marie Tooth Neuropathy Score-v2) ranges from 0-36. The disease severity is classified as mild (≤10), moderate (11 to 20), and severe (>21).
Changes from baseline in neurological examination at Weeks 1, 4, 12 and 24 | Weeks 1, 4, 12 and 24
  The principal investigator will assess the neurological examination which is investigated the evidence of muscle weakness in the arms, legs, hands, and feet; as well as signs of muscle wasting, reduced reflexes, and any sensory loss.
Changes from baseline in the overall neuropathy limitation scale (ONLS) at Weeks 4, 12 and 24 | Weeks 4, 12 and 24
  The Overall Neuropathy Limiting Scale (ONLS) assesses scale scores in the lower extremities as the Total Neuropathy Limiting Scale. A 1-point stage represents a clinically meaningful change in terms of disability.
Changes from baseline in functional disability using the functional disability scale (FDS) at Weeks 4, 12, and 24 | Weeks 4, 12, and 24
  The Functional Disability Scale (FDS) primarily evaluates impairment in motor function and is assessed by the neurologist (principal investigator) during the visit.
  The 9 stages of FDS are as follows:
  0; normal, 1; normal but with cramps and fatigability, 2; inability to run, 3; walking difficulty but still possible unaided, 4; If able to walk with a cane (walk with cane), 5; walk with crutches, 6; walk with a walker, 7; wheelchair bound, 8; bedridden.
Changes from baseline in the 10-meter walk test at Weeks 4, 12, and 24 | Weeks 4, 12, and 24
  This test measures the time required for a subject to walk 10 m through the 10-Meter Walking Test (10MWT)
Change from baseline in the fatty infiltration level of lower limb muscles at Week 24. | Week 24
  The degree of fat infilteration seen on MRI was classified into five grades from 0-4 and compared as follow: No fat infiltration at all (Grade 0; no fat), some traces of fat infiltration (Grade1; some fatty streak), more muscle than fat (Grade2; fat <muscle), when muscle and fat are similar (Grade3; fat = muscle), and when fat is more than muscle (Grade 4; fat>muscle).
Changes from baseline in the velocity of Motor and Sensory nerve conduction at Weeks 4, 12, and 24 | Weeks 4, 12, and 24
  Motor and sensory nerve conduction studies will be performed on the median nerve, ulnar nerve, peroneal nerve, tibial nerve, and sural nerve using skin surface stimulation electrodes and recording electrodes. using the skin surface stimulation and recording method.
  The studies will be performed with the amplitudes of the compound muscle action potential (CMAP) and the sensory nerve action potential (SNAP) from the positive maximum value to the negative maximum value.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical center, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No